CLINICAL TRIAL: NCT02226965
Title: A Phase II Study of PNT2258 in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: PNT2258 for Treatment of Patients With r/r DLBCL (Wolverine)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNT2258-03-DLBCL
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma, Diffuse Large B-Cell
Keywords: PNT2258; DLBCL; Diffuse Large B-cell Lymphoma; NHL; Non-Hodgkin's Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma | interventions — PNT100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PNT2258 (Experimental): PNT2258 will be administered at 120 mg/m2 on days 1-5 of a 21-day cycle. Treatment may continue unless there is disease progression or the occurrence of unacceptable toxicity for a total of 8 "induction" cycles of therapy. Subjects with CR/CMR, PR/PMR or SD/NMR at the end-of-cycle 8 scan then receive ongoing PNT2258 therapy at a dose of 100 mg/m2 on days 1-4 of a 28 day cycle until progressive disease, the occurrence of unacceptable toxicity, non-compliance, voluntary withdrawal or if in the opinion of the investigator the subject is no longer benefiting from exposure to PNT2258.
  Interventions: Drug: PNT2258

INTERVENTIONS:
Drug: PNT2258
  Other Names: DNAi, BCL2 targeted therapy

SUMMARY:
This study is sponsored by Sierra Oncology, Inc. formerly ProNAi Therapeutics, Inc. It is a multi-center, nonrandomized, open label, phase II investigation of PNT2258 to characterize anti-tumor activity and collect safety data on patients with relapsed or refractory (r/r) diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diffuse large B-cell lymphoma that is refractory to prior therapy or relapsed after prior therapy.

FDG PET-CT (disease) positive baseline scan with measurable disease.

The patient must have received prior therapy that included:

* CD20-targeted therapy (for example, rituximab),
* Alkylating agent (for example, cyclophosphomide), and
* Steroid, unless the patient is steroid intolerant

Exposure to at least 1 or 2 (but no more than 3) prior systemic cytotoxic chemotherapeutic regimens.

Note: Only those subjects who are not eligible for high-dose chemotherapy and autologous stem cell transplant (HD-ASCT), or who refuse HD-ASCT, are eligible with exposure to only 1 prior cytotoxic chemotherapeutic regimen.

ECOG performance status of 0-1.

The patient must be a stable baseline with CTCAE grade ≤ 2 regarding any acute or chronic toxicity associated with prior therapy, and have discontinued prior anti-cancer therapy for ≥ 14 days prior to C1D1; mitomycin-C for at least 6 weeks prior to C1D1; SCT ≥ 2 months prior to C1D1.

Note: Palliative steroids for control of disease-related symptoms are allowed and maintenance hormone therapy is allowed.

Adequate organ function including:

* Hematologic: ANC ≥ 0.5 x 10^9/L. and platelets ≥ 50 x 10^9/L.
* Hepatic: Total Bilirubin ≤ 2 x ULN (patients with Gilbert's syndrome must have total bilirubin ≤ 3 x ULN) and serum transaminase levels ≤ 2.5 x ULN. In the case of known liver metastasis (i.e., radiological or biopsy documented), serum transaminase levels must be ≤ 5 x ULN.
* Renal: Serum creatinine ≤ 2 x ULN, or creatinine clearance ≥ 60 mL/min/1.73 m2 for subjects with serum creatinine levels above 2 x ULN.

Willingness to: 1.) undergo pre-treatment biopsy to obtain adequate tissue for analysis (e.g., core needle, excisional or incisional tumor biopsy) or 2.) provide archived tumor (e.g., FFPE block) for analysis.

Exclusion Criteria:

Eligibility for high-dose chemotherapy (HDT) and stem cell transplant (SCT). Note: Subjects who progressed ≥ 2 months after HDT/SCT are eligible

Concurrent malignancies requiring treatment.

Primary mediastinal (thymic) large B-cell lymphoma

Symptomatic CNS or leptomeningeal involvement of lymphoma.

Concurrent clinically significant illness, medical condition, surgical history, physical finding, electrocardiogram or laboratory finding that, in the opinion of the investigator, could adversely affect the safety of the patient or impair the assessment of the study results.

Signs or symptoms of heart failure characterized as greater than NYHA Class II or other significant cardiac abnormalities.

Pregnant or breast-feeding.

Prior exposure to PNT2258.

Life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Klencke, MD, Study Chair — Sierra Oncology LLC - a GSK company
Locations (27):
- United States (26):
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of Southern California, Los Angeles, California
  - Colorado Blood and Cancer Institute, Denver, Colorado
  - Lynn Cancer Institute, Boca Raton, Florida
  - Bond Clinic, P.A., Winter Haven, Florida
  - Georgia Regents University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - UHC Oncology, Lafayette, Louisiana
  - Western Maryland Health System, Cumberland, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Michigan State University, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Bon Secours Saint Francis Cancer Center, Greenville, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Baylor Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Tyler Hematology Oncology, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia
  - Medical Oncology Associates, PS, Spokane, Washington
- Fundacion de Investigacion, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated in December 2014 and the first subject was enrolled on 10 December 2014. A total of 60 subjects were screened. Enrollment was closed as of 07 June 2016. Subjects were enrolled at oncology clinics in the USA.
Groups:
- PNT2258: PNT2258 was administered at a dose of 120 mg/m2, as a 3 - 4 hour intravenous (IV) infusion on days 1 through 5 of 21-day induction phase cycles (for eight cycles), followed by continuation phase therapy at a dose of 100 mg/m2, as a 2 - 3 hour intravenous (IV) infusion on days 1 through 4 of a 28-day cycle.
Period: Overall Study
Arm/Group | PNT2258
Started | 45
Completed (4 subjects completed the Induction Phase and 3 subjects started the Continuation Phase) | 4
Not Completed | 41

BASELINE CHARACTERISTICS:
Population: All patients who passed the screening in the study
Arm/Group | PNT2258
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 64 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The proportion of patients with complete response (CR/complete metabolic response [CMR]) or partial response (PR/partial metabolic response [PMR]) according to the revised 2014 International Working Group (IWG) criteria for lymphoma (Cheson 2014)
Time Frame: 19 months
Population: All enrolled population: All patients who passed the screening in the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PNT2258
Number analyzed (Participants) | 45
percentage of participants | 11.1 [3.7 to 24.1]

2. Secondary Outcome: Disease Control Rate
Description: The proportion of patients who have a response of stable disease (SD/no metabolic response [NMR]) or better by investigator assessment
Time Frame: 19 months
Population: All enrolled population: All patients who passed the screening in the study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PNT2258
Number analyzed (Participants) | 45
percentage of participants | 20.0 [9.6 to 34.6]

3. Secondary Outcome: Time to Response
Description: The number of months from Cycle 1 Day 1 until the date of the first documented response
Time Frame: 19 months
Population: All enrolled population: All patients who passed the screening in the study
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | PNT2258
Number analyzed (Participants) | 45
months | 2.2 [1.9 to 5.4]

4. Secondary Outcome: Progression-free Survival
Description: The number of months from C1D1 until the date of DLBCL progression or death from any cause, or to the last date at which progression status was adequately assessed for censored observation
Time Frame: 19 months
Population: All enrolled population: All patients who passed the screening in the study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PNT2258
Number analyzed (Participants) | 45
months | 1.9 [1.4 to 1.9]

5. Secondary Outcome: Safety - Assessment of Adverse Events
Description: Characterization of the type, frequency, severity, timing of onset, duration, and relationship to study drug of any treatment-emergent adverse events, laboratory abnormalities, serious adverse events or adverse events leading to discontinuation of study treatment
Time Frame: 36 months
Population: Safety population: All patients who received at least 1 dose of PNT2258
Measure: Number; unit: participants reporting at least 1 AE
Arm/Group | PNT2258
Number analyzed (Participants) | 45
participants reporting at least 1 AE | 45

6. Secondary Outcome: Overall Survival
Description: The number of months from C1D1 until the date of death from any cause, or to the last date at which survival status was adequately assessed for censored observations
Time Frame: 19 months
Population: All enrolled population: All patients who passed the screening in the study
Measure: Median (Full Range); unit: months
Arm/Group | PNT2258
Number analyzed (Participants) | 45
months | 9.8 [0.3 to 19.1]

7. Secondary Outcome: Duration of Overall Response
Description: The time from the initial CMR or PMR until the date of progression or death from any cause, or to the last date at which progression status was adequately assessed for censored observations
Time Frame: 19 months
Population: All enrolled population: All patients who passed the screening in the study
Measure: Median (Full Range); unit: months
Arm/Group | PNT2258
Number analyzed (Participants) | 45
months | 5.3 [0.0 to 8.3]

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events were collected until 30 days after the last dose of PNT2258 for each subject
Arm/Group | PNT2258
All-Cause Mortality (participants affected / at risk) | 11/45
Serious Adverse Events (participants affected / at risk) | 18/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PNT2258 (N=45)
Pyrexia (General disorders) | 5
Hypotension (Vascular disorders) | 3
Disease progression (General disorders) | 3
Sepsis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Cellulitis (Infections and infestations) | 1
Chills (General disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Septic shock (Infections and infestations) | 1
Spinal cord compression (Nervous system disorders) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PNT2258 (N=45)
Fatigue (General disorders) | 20
Nausea (Gastrointestinal disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 18
Pyrexia (General disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 13
Vomiting (Gastrointestinal disorders) | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 10
Decreased appetite (Metabolism and nutrition disorders) | 11
Dizziness (Nervous system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Constipation (Gastrointestinal disorders) | 10
Aspartate aminotransferase increased (Investigations) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Hypotension (Vascular disorders) | 8
Chills (General disorders) | 8
Alanine aminotransferase increased (Investigations) | 8
Insomnia (Psychiatric disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Hypoaesthesia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 5
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 5
Abdominal distension (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Hypertension (Vascular disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Sinus tachycardia (Cardiac disorders) | 4
White blood cell count decreased (Investigations) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Asthenia (General disorders) | 3
Blood creatinine increased (Investigations) | 3
Depression (Psychiatric disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Influenza like illness (General disorders) | 3
Lethargy (Nervous system disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Oedema peripheral (General disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes